CLINICAL TRIAL: NCT00061035
Title: A Phase 1, Evaluation of Transgenic Lymphocyte Immunization Vaccine in Subjects With Prostate Adenocarcinoma
Brief Title: Evaluation of Transgenic Lymphocyte Immunization Vaccine in Subjects With Prostate Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cosmo Bioscience (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLI-CA-TRT-001; NCT00066261 (obsolete NCT alias)
Record Dates: First submitted 2003-05-20; First posted 2003-05-22 (Estimated); Last update posted 2008-08-28 (Estimated); Status verified 2008-08

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Cancer; Immunotherapy
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Biological: Transgenic Lymphocyte Immunization Vaccine (TLI)

SUMMARY:
Dr. Frederick Millard, MD, Associate Clinical Professor at the UCSD Cancer Center, will be conducting a 12-week study in advanced prostate cancer patients. The study will be held at the UCSD Medical Center and will test an experimental investigational gene therapy vaccine designed to make the patient's immune system react against telomerase, an enzyme expressed in prostate cancer cells.

DETAILED DESCRIPTION:
The goal of the study is to determine the safety, feasibility, and tolerability of transgenic lymphocyte immunization (TLI). In this process patient's lymphocytes are rendered transgenic for a gene coding for selected portion of telomerase an enzyme expressed in the vast majority of cancer cells. Transgenic cells are then returned to the patient to produce an immune response targeted at cancer cells expressing telomerase. The Phase 1 trial will evaluate TLI in patients with advanced, androgen-independent prostate cancer with metastases confined to lymph nodes or bones.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, able to understand and sign the informed consent form.
* HLA-A2 positive.
* Expected survival ≥ 6 months.
* Histological evidence of adenocarcinoma of the prostate.
* (ECOG) Performance status 0, 1 or 2.

The following categories of subjects with androgen-independent prostate cancer are eligible:

* Progression of bidimensionally measurable disease assessed within 84 days (12 weeks) prior to enrollment.
* Progression of evaluable but not measurable disease (i.e., bone scan) assessed within 112 days (16 weeks) prior to enrollment.
* Rising PSA- Rising PSA is defined as at least two consecutive rises in PSA to be documented over a reference value (measure 1). The first rising PSA (measure 2) must be taken at least 7 days after the reference value. A third confirmatory PSA measure is required (2nd beyond the reference level) to be greater than the second measure, and it must be obtained at least 7 days after the 2nd measure. If this is not the case, a fourth PSA is required to be taken and be greater than the second measure. The subject must have a PSA ≥ 5 ng/ml in addition to increasing PSA to be eligible. No minimum PSA is required for subjects with measurable disease or non-PSA evaluable disease.
* All subjects must have had a CT scan of the abdomen and pelvis within 84 days (12 weeks) prior to enrollment.
* All subjects must also have had a bone scan within 112 days (16 weeks) prior to enrollment.
* Subjects must have been surgically or medically castrated. If method of castration is LHRH agonists (leuprolide or goserelin), then the subject should be willing to continue the use of LHRH agonists. Castration using LHRH agonist should not be interrupted and subjects who have stopped treatment should be willing to restart.
* If the subject has been treated with non-steroidal anti-androgens (flutamide, bicalutamide, nilutamide or ketoconazole), they must have been stopped at least 28 days prior to enrollment for flutamide or ketoconazole and at least 42 days prior to enrollment for bicalutamide or nilutamide and the subjects must have demonstrated progression.
* Subjects may have received prior surgery. However, at least 21 days must have elapsed since completion of surgery and subject must have recovered from all side effects.
* All subjects must have pre-study PSA within 28 days of enrollment.

Subjects must meet the following initial laboratory criteria:

* granulocytes ≥ 1500/ul
* platelet count ≥ 100,000/ul
* hemoglobin ≥ 10 gms/dl
* bilirubin ≤ 1.5 x ULN
* AST ≤ 1.5 x ULN
* Creatinine ≤ 1.5 x ULN
* Testosterone < 50ng/ml for those who have not had bilateral orchiectomy
* PSA ≥ 5ng/ml if no measurable disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2003-04

CONTACTS AND LOCATIONS:
Overall Officials: Frederick E. Millard, M.D, Principal Investigator — Associate Professor of Medicine at UCSD and Medical Director of the CTO of the UCSD Cancer Center
Locations (1):
- University of California, San Diego Cancer Center, San Diego, California, United States

REFERENCES:
- [Background] Zanetti M. Protocol #0207-545: a phase I/II, escalating dose, open-label evaluation of safety, feasibility, and tolerability of transgenic lymphocyte immunization (TLI) vaccine subjects with histologically proven prostate adenocarcinoma. Hum Gene Ther. 2003 Feb 10;14(3):301-2. No abstract available. PMID 12653092
- See also: Click here for more information about this study: Clinical Trial Vaccine Therapy for Prostate Cancer — http://cancer.ucsd.edu